CLINICAL TRIAL: NCT03505281
Title: Evaluation of a Functional Lymphocyte Test (QuantiFERON Monitor®) as a Prognostic Marker for Acute Community-acquired Pneumonia
Acronym: LYMPHONIE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BLOT 2017 LYMPHONIE
Record Dates: First submitted 2018-04-19; First posted 2018-04-23 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients
  Interventions: Biological: Blood samples
- Healthy volunteers
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — Patients:
  * 1 tube of 4 ml blood (Lithium Heparinate)
  * 3 tubes of 7 ml blood (EDTA)
  * 2 tubes of 7 ml blood (EDTA) for 20 NET Covid patients
  Healthy volunteers:
  * 1 tube of 4 ml blood (Lithium Heparinate)
  * 3 tubes of 7 ml of blood (EDTA)
  * 1 tube of 4 ml (citrate)

SUMMARY:
Lower respiratory infections, or pneumonia, remain the third leading cause of death worldwide, despite progress in vaccinating at-risk populations and improved resuscitation techniques.

Research shows that immune defences are weakened during severe infections. This immune weakening could alter resistance to bacterial infection and facilitate death, but also facilitate the onset of secondary infections.

Through this study, investigators wish to evaluate a biomedical test (derived from a blood sample - Quantiferon Monitor test), aimed at measuring the immune response of certain immune cells (lymphocytes).

The objective of the study is to determine whether this test can predict the occurrence of death during pneumonia.

If this hypothesis is verified, it would make it possible to use this test as a marker to identify patients at risk of death, and would open up new therapeutic prospects in order to provide patients with severe pneumonia with a treatment that stimulates their immune defences.

Recently, COVID-19 has changed the epidemiology and management of acute community-acquired pneumonia. Numerous studies, including some recently published ancillary studies of the Lymphony study, suggest that a deregulated immune response could contribute to the poor patient prognosis. Different determinants could contribute to this. Endotoxemia reflects the elevation of plasma LPS concentrations and represents a major Gram-negative determinant. Endotoxemia also seems to be observed during infectious pneumopathies, even though the main causative agents are devoid of LPS. The genesis of this endotoxemia and its intensity could reflect a digestive bacterial translocation phenomena that is correlated with severity.

Concerning the secondary objectives of the COVITOXEMIA ancillary study: the main hypothesis is that severe pneumopathies related to SARS-CoV2- are associated with endotoxemia.

Furthermore, early work comparing the immune response during severe SARS-CoV-2-related lung disease to immune responses of other origins demonstrated higher concentrations of CXCL10, GM-CSF, and VCAM1 during COVID-19. Since these 3 markers mediate activation (GM-CSF), chemotaxis (CXCL10), and diapedesis (VCAM-1) of myeloid cells, these results suggest an important role for their activation during COVID-19, especially of neutrophils.

Regarding the secondary objectives of the NETCovid study:

In an attempt to better characterize the specific pathogenesis of COVID-19, which contributes to the poor outcome, the objective is to compare the neutrophil immune response between patients with and without SARS-CoV-2 related severe pneumonia, considering the levels of biomarkers of activation (including NETose), degranulation and chemotaxis of neutrophils.

ELIGIBILITY:
Inclusion Criteria:

GROUP OF PATIENTS WITH PNEUMONIA

* Patient with acute pneumonitis:

  1) Acute signs and symptoms of lung disease (new or worsening), including at least 2 of the following:
* Cough
* Dyspnea
* Purulent sputum
* Chest pain
* Temperature ≥ 38°C or < 35°C 2) and new radiological pulmonary infiltrate (X-ray or CT scan on admission)
* Community Acquired Pneumonia:
* Pneumonia present on admission or diagnosed within 48 hours of admission,
* Poor prognosis according to the new quick SOFA sepsis score; poor prognosis is defined if at least 2 of the following criteria are present:
* Systolic blood pressure ≤ 100 mm Hg,
* Respiratory rate ≥ 22,
* Altered consciousness (Glasgow score < 15). And/or need for mechanical ventilation (invasive or non-invasive). And/or need for use of vasopressors for hemodynamic failure.
* Patient of legal age who has given informed consent
* Patient affiliated to the national health insurance system
* For patients with "severe SARS-CoV-2 pneumonia":

  1. Respiratory specimen positive for SARS-CoV-2 (PCR)
  2. And without Gram-negative bacilli found on respiratory and blood samples.

CONTROL GROUP (HEALTHY VOLUNTEERS):

* No infection in the previous or current 30 days

  1. No fever reported in the previous 30 days
  2. No antibiotics taken in the previous 30 days
  3. Temperature < 37.8°C on the day of inclusion
  4. Absence of clinically suspected infection
* No surgery in the previous 30 days
* Patient over 18 years of age who has provided informed consent
* Patient affiliated to the national health insurance system

Exclusion Criteria:

* Person protected by law
* Minor
* Pregnant, parturient or breastfeeding woman
* Patient with a known primary or secondary immune deficiency (radiation therapy, chemotherapy, immunosuppressive therapy or systemic corticosteroid therapy (> 0.15 mg/kg/day of prednisone equivalent for more than 2 weeks or "bolus" higher than 2 mg/kg/day of prednisone equivalent in the 3 months prior to inclusion), HIV infection, primary cellular immune deficiency)
* Presenting a chronic disorder known to cause deep lymphopenia (Cirrhosis, lympho or myeloproliferative syndrome, solid cancer or active systemic lupus erythematosus) and/or a condition known to cause a substantial increase in INF-γ (active hepatitis B)
* Patient who was hospitalized in the 3 months prior to inclusion for sepsis according to the new SOFA quick criteria
* Decision to limit care
* Treatment with Interferon initiated prior to study sampling

EXCLUSION CRITERIA

* For the pneumopathy group: Failure to take a sample for the QFM within 48 hours of admission.
* For the control group: CRP greater than 15 mg/L at the time of sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute community-acquired pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Death | 30 days following hospitalization for community-acquired pneumonia

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blot M, de Maistre E, Bourredjem A, Quenot JP, Nguyen M, Bouhemad B, Charles PE, Binquet C, Piroth L. Specific Features of the Coagulopathy Signature in Severe COVID-19 Pneumonia. Front Med (Lausanne). 2021 Aug 4;8:675191. doi: 10.3389/fmed.2021.675191. eCollection 2021. PMID 34422854
- [Derived] Blot M, David Masson, Nguyen M, Bourredjem A; LYMPHONIE Study Group; Binquet C, Piroth L. Are adipokines the missing link between obesity, immune response, and outcomes in severe COVID-19? Int J Obes (Lond). 2021 Sep;45(9):2126-2131. doi: 10.1038/s41366-021-00868-5. Epub 2021 May 31. PMID 34059786
- [Derived] Blot M, Bour JB, Quenot JP, Bourredjem A, Nguyen M, Guy J, Monier S, Georges M, Large A, Dargent A, Guilhem A, Mouries-Martin S, Barben J, Bouhemad B, Charles PE, Chavanet P, Binquet C, Piroth L; LYMPHONIE study group. The dysregulated innate immune response in severe COVID-19 pneumonia that could drive poorer outcome. J Transl Med. 2020 Dec 3;18(1):457. doi: 10.1186/s12967-020-02646-9. PMID 33272291